CLINICAL TRIAL: NCT06614790
Title: Patient Outcomes and Safety of Niraparib as Maintenance Treatment in Patients With Newly Diagnosed Advanced Platinum- Sensitive, Ovarian Cancer. The First Real-World Evidence Study From Poland.
Brief Title: Niraparib Maintenance Treatment in Patients With Newly Diagnosed Advanced Platinum- Sensitive, OC. The First Poland RWE Study.
Acronym: NIRAPARIB
Status: Recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: NIRAPARIB; GSK (Other: ID 15146)
Record Dates: First submitted 2024-09-13; First posted 2024-09-26 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer
Keywords: maintenance treatment; iPARP; advanced ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with advanced, high-grade ovarian cancer who respond on the first line therapy (NED, CR,PR)
  Interventions: Drug: Niraparib 200/300 MG

INTERVENTIONS:
Drug: Niraparib 200/300 MG — We expect to enroll approximately 300 patients from about 10 sites. Treatment part of study.
  Part I- looking retrospectively at the time period JAN 2021-MAR 2023. The retrospective data will include patients who are enrolled in niraparib treatment:
  * under the EAP (started in JAN 2021, in continuation)
  * under the B.50 drug program, which began in January 2022 Of note, the retrospective multi-center observational study will involve about 30 patients treated with niraparib in EAP (FIGO III R0 after PDS included) and patients who were treated with niraparib before starting RWE (about 120 pts) (JAN 2021- MAR 2023) by the drug program B.50 which has been started to adapt on 1st of Jan, 2022.
  FIGO III PDS to R0 patients are included to this study. Part II- looking prospectively at the time period APR 2023 to DEC 2025. The prospective data will include patients who are enrolled in niraparib treatment under the B.50 drug program.
  The prospective multi-center observational study will i

SUMMARY:
The study is observational, not interventional. The study will include patients with advanced ovarian cancer who have been treated in Poland based on a previous early access program, and who are currently being treated under the B.50 drug program, funded by the National Health Fund.

Only patients currently being treated in the B.50 program at 10 selected centers listed on this site may be included in the study.

Of course, any patient in Poland eligible for maintenance treatment with niraparib can receive the drug, regardless of participation in this RWE study.The treatment involves administering niraparib as maintenance therapy for 3 years after the completion of chemotherapy, provided that the patient has responded to systemic treatment (NED, CR, PR).

DETAILED DESCRIPTION:
Although over the last 2 decades the surgical management of ovarian cancer has improved with more chemotherapy options are available, however 5-year survival rates have remained relatively stable at 25 to 40% (36) The proposed real-life observation study can deliver valuable real-world information about niraparib patient outcomes and safety complementing the results of the PRIMA and PRIME clinical trials. This will also include establishing the importance of KELIM as a predictor of maintenance therapy choices. The multicenter design of the study will allow collection of data from a relatively large and representative group of patients within the Polish Drug program B.50. To this time, no study has been published about niraparib patient outcomes and safety in Poland.

This study will also include evaluation of patient outcomes when initiating therapy up to 4, 8, 12 weeks after completion of platinum based chemotherapy.

The population of patients included in the study will come from two programs: EAP and B.50.

EAP is an early access program sponsored by GSK, which has been operating in Poland since 2021 Jan. The inclusion criteria for EAP contained the same measurable parameters as the B.50 drug program offers.

The B.50 drug program is a ministerial program guaranteeing the Polish patients with advanced ovarian cancer access to approved medicines like maintenance treatment with PARP inhibitors, including niraparib.

The B.50 and EAP inclusion criteria are in accordance with the study protocol.

Primary Objective

* Primary objectives will be to describe patient and disease characteristics for patients receiving niraparib treatment in Poland.
* To quantify PFS: the primary PFS analysis will be based upon the Investigator's assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria, Appendix 2. The day considered as disease progression is the day of the CT examination on which progression was found according to RECIST 1.1 criteria
* PFS measured from the time of the first dose of niraparib.
* Primary objectives will also estimate safety and tolerability of niraparib treatment in Poland. Strict monitoring of safety profile (e.g. blood test is performed every 7 days during first month of treatment and after each changing of dose, blood pressure is performed every 7 days within the first two months then every month within the first year).

Secondary Objectives

* OS (Overall Survival)
* Chemosensitivity based on KELIM as a surrogate marker for platinum sensitivity to assess for niraparib response as a standard procedure due to the B.50 drug program
* Evaluation of outcomes of including patients in therapy up to 4, 8, 12 weeks after completion of platinum-based chemotherapy
* TFST (Time to the First Subsequent Therapy)
* DCR (Disease Control Rate).

INVESTIGATIONAL PLAN

Overall Study Design Patients who complete the Chemotherapy Treatment Period without progressive disease (CR, PR, NED) will start Maintenance Treatment with niraparib after Cycle 6 up to 12 weeks after completion of the chemotherapy.

Prior to receiving oral maintenance treatment, patients must have a CBC that demonstrates adequate recovery from hematologic toxicity from chemotherapy:

* Absolute neutrophil count ≥1,500 cells/μL
* Platelet count ≥100,000 cells/μL
* Hemoglobin ≥10 g/dl

Number of Patients and Study Design We expect to enroll approximately 300 patients from about 10 sites. Treatment part of study.

Part I- looking retrospectively at the time period JAN 2021-MAR 2023. The retrospective data will include patients who are enrolled in niraparib treatment:

* under the EAP (started in JAN 2021, in continuation)
* under the B.50 drug program, which began in January 2022 Of note, the retrospective multi-center observational study will involve about 30 patients treated with niraparib in EAP (FIGO III R0 after PDS included) and patients who were treated with niraparib before starting RWE (about 120 pts) (JAN 2021- MAR 2023) by the drug program B.50 which has been started to adapt on 1st of Jan, 2022.

FIGO III PDS to R0 patients are included to this study. Part II- looking prospectively at the time period APR 2023 to DEC 2025. The prospective data will include patients who are enrolled in niraparib treatment under the B.50 drug program.

The prospective multi-center observational study will involve about 150 patients with ovarian cancer (OC) who have been treated in about 10 OC gyn- oncocenters in Poland (OCgoC) (APR 2023- DEC 2025).

Study follow up Part III- survival follow up after treatment part of study (from JAN 2026 - DEC 2026).

Chemotherapy Treatment Period Not covered by the study protocol.

Maintenance Treatment Period All the patients will be given a sequential number by the system. Additionally, each patient from the EAP will have individual number which was given to them. In the CRF there will be additional information that there is a patient in the EAP phase of the study. Patients who have responded to first-line chemotherapy (NED, CR, PR) and with recovery to baseline of any hematologic toxicities will enter the Maintenance Treatment Period. Oral niraparib will be dispensed to patients on Day 1 of every 28-day cycle beginning with Cycle 1 of the Maintenance Treatment Period for up to 3 years in the absence of PD, unacceptable toxicity, or patient withdrawal, or based on Investigator's decision.

The recommended dose is 200 mg per day (2 capsules). Patients with a baseline body weight of ≥77 kg and baseline platelet count of ≥150,000 cells/μL will take 3 capsules of 100 mg strength (300 mg/day) at each dose administration.

Dose modifications will not be based upon changes in the patient's actual body weight during their study participation.

The inclusion criteria, the way of monitoring, both in a prospective and a retrospective cohort, will be followed by the B.50 drug program criteria. For that reason CA125 measurements necessary for KELIM as well as RECIST data are available in both cohorts during the whole period of time.

Duration of Treatment Patients may continue niraparib treatment for up to 3 years according to the B.50 drug program.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female, ≥18 years of age, able to understand the study procedures, and agree to participate in the study by providing written informed consent.
2. Patients with a histologically confirmed diagnosis of nonmucinous high - grade epithelial ovarian cancer (serous, endometrial) that is stage III or IV according to the FIGO criteria.
3. All patients with Stage IV disease are eligible. This includes those with inoperable disease, those who undergo PDS (R0 or macroscopic disease), or those for whom NACT is planned.
4. Patients with Stage III are eligible if they meet the following criteria:

   1. All FIGO III patients in spite of residual disease and cytoreductive surgery.
   2. All patients with inoperable Stage III disease.
   3. All Stage III patients after NACT chemotherapy.
5. FFPE tumor tissue sample must be available for molecular analysis.
6. Patients of childbearing potential must have a negative serum or urine pregnancy test (beta human chorionic gonadotropin) within 72 hours prior to receiving the first dose of study treatment.
7. Patients must be postmenopausal, free from menses for >1 year, surgically sterilized, or willing to use highly effective contraception to prevent pregnancy (see 0) or must agree to abstain from activities that could result in pregnancy throughout the study, starting with enrollment through 180 days after the last dose of study treatment.

   1. Serum creatinine ≤1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault equation
   2. Total bilirubin ≤1.5 × ULN or direct bilirubin ≤1.5 × ULN
   3. AST and ALT ≤2.5 × ULN unless liver metastases are present, in which case they must be ≤5 × ULN
8. Patients must have an ECOG score of 0 or 1.
9. Patients must have normal BP or adequately treated and controlled hypertension.
10. Patients must be able to take oral medication.

Exclusion Criteria:

1. Patient has mucinous, germ cell, transitional cell, or undifferentiated tumor.
2. Patient has low-grade or Grade 1 epithelial ovarian cancer.
3. Patient has a known condition, therapy, or laboratory abnormality that might confound the study results or interfere with the patient's participation for the full duration of the study treatment in the opinion of the Investigator.
4. Patient is pregnant or is expecting to conceive children while receiving study drug or for up to 180 days after the last dose of study drug. Patient is breastfeeding or is expecting to breastfeed within 30 days of receiving the final dose of study drug (women should not breastfeed or store breastmilk for use, during niraparib treatment and for 30 days after receiving the final dose of study treatment).
5. Patient has any known history or current diagnosis of MDS or AML.
6. Hypersensitivity to the active substance or to any of the excipients including tartrazine.
7. Hypertension-Participants have systolic BP >140 mmHg or diastolic BP >90 mmHg that has not been adequately treated or controlled.
8. Patients with prior history of PRES.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who complete the Chemotherapy Treatment Period without progressive disease (CR, PR, NED) will start Maintenance Treatment with niraparib after Cycle 6 up to 12 weeks after completion of the chemotherapy.
  Prior to receiving oral maintenance treatment, patients must have a CBC that demonstrates adequate recovery from hematologic toxicity from chemotherapy:
  * Absolute neutrophil count ≥1,500 cells/μL
  * Platelet count ≥100,000 cells/μL
  * Hemoglobin ≥10 g/dl
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability. | 27 months
  Safety and tolerability of niraparib treatment in Poland. Strict monitoring of safety profile (e.g. blood test is performed every 7 days during first month of treatment and after each changing of dose, blood pressure is performed every 7 days within the first two months then every month within the first year).
PFS measured from the time of the first dose of niraparib. | 48 months
  The primary PFS analysis will be based upon the Investigator's assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria, Appendix 2. The day considered as disease progression is the day of the CT examination on which progression was found according to RECIST 1.1 criteria. PFS is defined as the time from first dose of niraparib starting until objective tumor progression or death.

SECONDARY OUTCOMES:
Chemosensitivity based on KELIM. | 100 days
  Chemosensitivity based on KELIM as a surrogate marker for platinum sensitivity to assess for niraparib response as a standard procedure due to the B.50 drug program.I will be measured after the chemotherapy based on CA125 making during the first 100 days of treatment.
OS (Overall Survival). | 48 months
  Overall survival is defined as the time from the start of therapy to the day of patient's death to any cause.
PFS depending on starting niraparib therapy. | 48 months
  Evaluation of outcomes of including patients in therapy up to 4, 8, 12 weeks after completion of platinum-based chemotherapy
DCR (Disease Control Rate). | 48 months
  Disease control rate (DCR) is defined as the percentage of patients who have achieved complete response, partial response, and stable disease to the niraparib intervention.
TFST (Time to the First Subsequent Therapy). | 48 months
  TFST is defined as the time from initiation of first-line chemotherapy until the start of subsequent therapy or death.

CONTACTS AND LOCATIONS:
Locations (11):
- Poland (11):
  - Oddział Onkologii Ginekologicznej Białostockiego Centrum Onkologii, Bialystok
  - Klinika Położnictwa i Ginekologii, Ginekologii Onkologicznej Uniwersyteckie Centrum Kliniczne, Gdansk
  - III Klinika Radioterapii i Chemioterapii Narodowego Instytutu Onkologicznego w Gliwicach, Gliwice
  - Świętokrzyskie Centrum Onkologii, Kielce
  - Klinika Ginekologii Onkologicznej Narodowego Instytutu Onkologicznego w Krakowie, Krakow
  - I Katedra i Klinika Ginekologii Onkologicznej i Ginekologii Uniwersytetu Medycznego w Lublinie, Lublin
  - Opolskie Centrum Onkologii, Opole
  - Oddział Onkologii Klinicznej i Radioterapii, Siedleckie Centrum Onkologii, Siedlce
  - Klinika Ginekologii Operacyjnej i Onkologii Ginekologicznej Dorosłych i Dziewcząt PUM, Szczecin
  - , Klinika Ginekologii Onkologicznej, Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie w Warszawie, Warsaw
  - Klinika Ginekologii Onkologicznej, Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie w Warszawie, Warsaw